CLINICAL TRIAL: NCT06276881
Title: Pain Relief Through Artificial Intelligence (AI) -Guided Dynamic Neuromodulation
Brief Title: Visual Stimulation for Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dandelion Science (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DSC1001; 1R43DA054845-01 (NIH)
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Photic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Controls (Experimental)
  Interventions: Behavioral: Visual Stimulation

INTERVENTIONS:
Behavioral: Visual Stimulation — AI-guided visual stimuli presented on an electronic screen

SUMMARY:
The goal of this study is to investigate a novel neuromodulatory approach utilizing visual stimulation to impact pain perception in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes
* Participants of diverse ethnic and racial backgrounds
* Participants who speak, read, and understand English and are willing and able to provide written informed
* 18 to 50 years old

Exclusion Criteria:

* Participants with neurologic, endocrine, renal, gastrointestinal, and chronic pain disease
* Participants who use unprescribed drugs or medications
* Chronically medicated participants
* Participants with photosensitivity and epileptic seizures
* Participants who have undergone major surgery within two months of the experiment date
* Participants with cardiac disorders
* Participants who are pregnant
* Prisoners
* Participants who are unable to provide consent
* Participants diagnosed with a psychiatric disorder that is likely to interfere with the conduct of the study
* Participants with implanted electronic devices of any kind, including pace-makers, electronic infusion pumps, stimulators, defibrillators

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Executive Officer (CEO), Principal Investigator — Dandelion Science Corp
Locations (1):
- Dandelion Science, Hoboken, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Visual Stimulation: AI (Artificial-Intelligence)-guided visual stimuli presented on an electronic screen
Period: Overall Study
Arm/Group | Healthy Controls
Started | 75
Generating and Validating the Stimuli | 10
Testing Medoc, Validating Thermal Responses | 18
Testing Pain Relief (Analysis Group) | 47
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Controls
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.97 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Score
Description: Standard computerized scale of perceived pain level. The scale ranges from 0 to 100, a score of "0" indicating "No Pain" and a score of "100" indicating "Most Pain". Higher score indicates a worse outcome as perceived pain is increasing, lower score indicates a better outcome as perceived pain is decreasing.
Time Frame: Up to 2 hours
Population: Sixteen participants removed from analysis due to noisy data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
score on a scale
  VAS Score in Response to No Visual Stimulation | 24.77 (20.51)
  VAS Score in Response to Flicker Visual Stimulation | 25.02 (21.55)
  VAS Score in Response to Abstract Visual Stimulation | 25.19 (21.13)
  VAS Score in Response to Semantic Visual Stimulation | 23.64 (21.19)
Statistical Analysis 1: Comparison: Healthy Controls; Test type: Superiority; p = .37, t-test, 1 sided; Multiple regression analysis

2. Primary Outcome: Event-related Potential (ERP)
Description: Evoked event-related neural response to contact heat perception measured by EEG (electroencephalography), P300 component
Time Frame: Up to 2 hours
Population: Sixteen participants' data removed due to noisy data
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Controls
Number analyzed (Participants) | 31
Participants | 31
Statistical Analysis 1: Comparison: Healthy Controls; Test type: Superiority; p = .07, ANOVA

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT06276881/Prot_SAP_000.pdf